CLINICAL TRIAL: NCT06028074
Title: A First-in-Human, Open-Label, Phase 1/2 Dose-Escalation With Enrichment and Dose-Expansion Study to Investigate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Antitumor Activity of GIM-122 as a Single Agent in Adult Subjects With Advanced Solid Malignancies
Brief Title: Safety and Tolerability Study of GIM-122 in Subjects With Advanced Solid Malignancies
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Georgiamune Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIM122-CT01
Record Dates: First submitted 2023-08-31; First posted 2023-09-07 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Advanced Solid Malignancies
Keywords: solid tumor; advanced malignancies; GIM-122

STUDY DESIGN:
Intervention Model Description: Part A: Dose Escalation and Enrichment, Part B: Dose Expansion in specified tumor types
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Intravenous administration of GIM-122 (Experimental): GIM-122
  Interventions: Drug: GIM122

INTERVENTIONS:
Drug: GIM122 — GIM-122 administered IV once every 3 weeks or every 2 weeks
  Other Names: GIM-122

SUMMARY:
GIM-122 is a first-in-class, humanized immunoglobulin G1 kappa dual functioning monoclonal antibody (DFA). This phase 1 / 2 study plans to evaluate the safety, tolerability, pharmacokinetics and clinical efficacy of intravenous (IV) administration of GIM-122 in adults with advanced malignancies.

DETAILED DESCRIPTION:
This is a Phase 1/2, open label, first-in-human (FIH), multicenter, dose escalation study with enrichments and dose expansion cohorts at RP2D, designed to evaluate the safety, tolerability, PK, pharmacodynamics, and preliminary antitumor activity of GIM-122 administered as a single agent in adults with advanced solid malignancies. This study will be conducted in 2 parts: Phase 1 or Part A (dose escalation and enrichment) and Phase 2 or Part B (dose optimization and cohort expansion).

ELIGIBILITY:
Inclusion Criteria:

General

* Written informed consent
* ECOG performance status 0-1.
* Laboratory assessment 28 days prior to enrollment for assessment of acceptable cardiac, renal and hepatic functions
* Recommended Double methods of contraception 90-days post treatment Cancer Specific
* Histologically or cytologically confirmed locally advanced/unresectable or metastatic solid tumor
* Received FDA approved treatment of PD-1 inhibitor or PD-L1 inhibitor for advance malignant tumors and have progressed/relapsed, are refractory, or intolerant
* Measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1
* Had prior therapy with PD-1/PD-L1 inhibitors. Other checkpoint inhibitors (ie, CTLA4, LAG3) are permitted if they did not lead to treatment discontinuation
* No other lines of therapy that are available

Exclusion Criteria:

General

* Enrolled in any other interventional clinical trial, starting within 4 weeks of the first dose of GIM-122 and throughout the duration of the study, or is receiving other therapy directed at their malignancy
* Women who are pregnant or breastfeeding
* History of cardiac issues, pulmonary embolism, active and clinically significant bacterial, fungal, or viral infection ≤ 6 months prior to dosing
* Contraindications to the imaging assessments or other study procedures that subjects will undergo or any medical or social condition that, in the opinion of the investigator, might place a subject at an increased risk, affect compliance, or confound safety or other clinical study data interpretation Cancer Specific
* Current second malignancy at other sites
* Leptomeningeal disease
* Spinal cord compression
* Symptomatic or new or enlarging central nervous system (CNS) metastases

Treatment-specific Exclusion Criteria

* Ongoing toxicity > Grade 1 from prior therapy according to Common Terminology Criteria for Adverse Events (CTCAE) v 5.0
* Has undergone a major surgery < 1 month prior to administration of GIM-122
* Has received radiation therapy within 2 weeks prior to administration of GIM-122
* Has undergone or is anticipated to undergo organ transplantation including allogeneic or autologous stem cell transplantation at any time
* Has received systemic anti-cancer therapy within 2 weeks and cytotoxic agents that have a major delayed toxicity within 4 weeks, of the first dose of GIM-122
* Prior treatment with other immune modulating agents within < 4 weeks prior to the first dose of GIM-122.
* Has a diagnosis of immunodeficiency, either primary or acquired
* Has received treatment with systemic steroids or any form of immunosuppressive therapy within 14 days prior to administration of GIM-122
* Has active or prior history of autoimmune disease, including ulcerative colitis and Crohn's disease, or any condition that requires systemic steroids.
* Has a known severe intolerance to or hypersensitivity reactions to monoclonal antibodies, Fc-bearing proteins, or IV immunoglobulin preparations; prior history of human anti-human antibody response; known allergy to any of the study medications, or excipients in the various formulations of any agent.
* Has received live vaccines within 30 days of study initiation (inactivated vaccines are allowed; seasonal vaccines should be up to date > 30 days prior to administration of GIM-122).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicities [DLT] with GIM-122 | 18 months
  To identify dose limiting toxicities [DLT] with GIM-122
Maximum tolerated dose [MTD] of GIM-122 | 18 months
  To identify maximum tolerated dose [MTD] of GIM-122
Recommended Phase 2 Dose [RP2D] of GIM-122 | 18 Months
  To identify Recommended Phase 2 Dose [RP2D] of GIM-122
Overall response rate (ORR) -Part B of the study | 36 months
  To identify overall response rate (ORR) in patients with advanced malignant tumors who are refractory/ resistant to PD-1 and PD-L1 therapy
Anti-tumor activity of GIM-122 | 36 months
  To assess anti-tumor activity of GIM-122 as a single agent in patients with advanced malignant tumors who are refractory/ resistant to PD-1 and PD-L1 therapy
Incidence and severity of AE / SAEs and tolerability | 36 months
  To assess incidence and severity of AE / SAEs and tolerability assessed by CTCAE grading

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) | 36 months
  To preliminarily evaluate the AUC in patients with advanced malignant tumors
Peak Plasma Concentration (Cmax) | 36 months
  To preliminarily evaluate Cmax in patients with advanced malignant tumors
Time of peak plasma concentration (Tmax) | 36 months
  To preliminarily evaluate Tmax in patients with advanced malignant tumors
Overall Response Rate (ORR) - Part A of the study | 36 months
  To preliminarily evaluate ORR in patients with advanced malignant tumors
Duration of response (DOR) | 36 months
  To preliminarily evaluate DOR in patients with advanced malignant tumors
Disease control rate (DCR) | 36 months
  To preliminarily evaluate DCR in patients with advanced malignant tumors
Best overall response (BOR) | 36 months
  To preliminarily evaluate BOR in patients with advanced malignant tumors
Progression-free survival (PFS) | 36 months
  To preliminarily evaluate PFS in patients with advanced malignant tumors
Overall survival (OS) rates at 12 months | 36 months
  To preliminarily evaluate OS in patients with advanced malignant tumors at 12 Months
Tumor expression of immunological markers | 36 months
  To analyze tumor expression of immunological markers

CONTACTS AND LOCATIONS:
Overall Officials: Omid Hamid, MD, Principal Investigator — The Angeles Clinic and Research Institute
Locations (11):
- United States (11):
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - UCLA Hematology/Oncology, Los Angeles, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Florida Cancer Specialists, Sarasota, Florida
  - Norton Cancer Institute, Louisville, Kentucky
  - Rutgers Cancer Institute of NJ, New Brunswick, New Jersey
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Texas Oncology - Baylor Sammons Cancer Center, Dallas, Texas
  - NEXT Oncology Dallas, Irving, Texas
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No